CLINICAL TRIAL: NCT05671458
Title: Multiparametric Imaging-based Intraoperative Navigation for Guidance of Surgical Resection and Postoperative Radiotherapy in Patients With Head-and-neck Tumors - NAVIGATORR
Brief Title: Multiparametric Imaging-based Intraoperative Navigation for Guidance of Surgical Resection and Postoperative Radiotherapy in Patients With Head-and-neck Tumors
Acronym: NAVIGATORR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juergen Debus (Other)
Responsible Party: Sponsor-Investigator, Juergen Debus, PD Dr. Sebastian Regnery, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAVIGATORR
Record Dates: First submitted 2022-12-16; First posted 2023-01-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Tumors
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: intraoperative navigation and creation of tumor resection maps — TRM are based on intraoperative navigation data and yield anatomically accurate marks of the tumor resection margin and potential residual tumor areas on clinical imaging. These marks will be annotated with histopathological information. Subsequently, the resulting 3-dimensional TRM will be imported into the radiotherapy planning system as part of a multidisciplinary workflow.

SUMMARY:
The overarching goal of the NAVIGATORR trial is the improvement of local tumor control in head-and-neck cancer (HNC) by increasing the precision of surgical resection and individualization of radiotherapy. Squamous cell carcinomas (SCC) together with salivary gland carcinomas (adenoid cysytic Carcinoma (ACC), mucoepidermoid Carcinoma (MEC), adenocarcinoma (AC)) represent the most common entities in German head and neck oncology. In localized tumors, primary tumor resection with possible adjuvant (chemo)radiotherapy is still the treatment of choice. Advances in targeted therapy and immunotherapy have greatly expanded the repertoire of medical oncology in recent years. In particular, prognosis of patients with end-stage non-small cell lung cancer (NSCLC) has been improved and even patients with advanced head and neck disease can be offered new second line regimes. Importantly, all of these advances are based on personalized and targeted therapies. Unfortunately, surgical oncology in the head-and-neck region has not yet shown such developments towards individualized treatment, so that the rates of safe oncological resections (clear resection margins) haven been stagnating. Despite advances in reconstructive surgery that allow the resection of head-and-neck tumors that would not have been operable 10 - 15 years ago, the basic principles of the resection margin and especially margin evaluation have remained unchanged. The technique of navigation-based tumor resection and the annotation of biopsies by titanium clip-markings or special annotation have been described, but only in small case series and without proving the benefit of the method concerning clinically relevant parameters.

Therefore, the NAVIGATORR trial will enroll 60 patients with HNC of the midface that will undergo navigation-based surgery. Importantly, interdisciplinary data exchange of the intraoperative navigation data between surgeons, pathologists and radiation oncologists will be established. Clear surgical margins (distance between tumor cells and resection border > 5 mm) have been defined as primary endpoint. Secondary endpoints such as dosimetric assessment of individualized radiotherapy plans, local tumor control or overall survival should then be compared to data from the literature to further assess this multidisciplinary approach.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a malignancy (squamous cell carcinoma (SCC), adenocarcinoma (AC), mucoepidermoid carcinoma (MEC), adenoidcystic carcinoma (ACC)) of the midface, upper jaw and skull-base (e.g. based on imaging-studies and/or biopsies)
* Indication of surgical tumor resection according to multidisciplinary tumor conference
* Probably indication for postoperative radiotherapy (e.g. T3/4 tumor)
* Medical operability and written informed consent of the patient to undergo surgical resection (as indicated clinically)
* Patient age ≥ 18 years
* Karnofsky performance index ≥ 60%
* For women with childbearing potential: adequate contraception
* Ability of subject to understand character and individual consequences of the trial
* Written informed consent to participate in this trial

Exclusion Criteria:

* Contraindications against radiotherapy, especially pregnant or lactating women
* Refusal of the patient to take part in the study
* Participation in another competing clinical study or observation period of competing trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety of tumor resection | within 24 month after radiotherapy
  occurence of clear resection margins according to NCCN guidelines.

SECONDARY OUTCOMES:
local tumor control | within 24 month after radiotherapy
  Local progression is defined as progressive disease at the original tumor site according to the Response Evaluation Criteria in Solid Tumors (RECIST) in the current version 1.1.

OTHER OUTCOMES:
distant tumor control | within 24 month after radiotherapy
  Distant progression is defined as progressive disease according to RECIST v1.1 outside the original tumor site
Progression-free survival | within 24 month after radiotherapy
  Progression-free survival is defined as the time interval from surgical resection until the day of a progressive disease according to RECIST v1.1 at any site or death of any cause
Overall survival | within 24 month after radiotherapy
  Overall survival is defined as the time interval from surgical resection until death
Treatment-related toxicity | within 24 month after radiotherapy
  Treatment-related side effects will be assessed clinically and radiographically according to the CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy, University of Heidelberg, Heidelberg, Germany